CLINICAL TRIAL: NCT06443580
Title: The Relationship Between Interoception and Psychological Outcomes: A Mind-Body Intervention in Patients With Pulmonary Hypertension
Brief Title: Interoceptive Intervention for Pulmonary Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Principal Investigator, Derick Moore, Trainee Clinical Psychologist, Golden Jubilee National Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/MISC/01
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Interoception; Pulmonary Hypertension
Keywords: interoception; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group based interoceptive intervention (Experimental): an 8 week online group intervention where participants will learn skills to improve interoception and connect with their body.
  Interventions: Other: interoceptive group based intervention
- waitlist (No Intervention): participants will wait until first group have completed intervention before commencing themselves

INTERVENTIONS:
Other: interoceptive group based intervention — 8 week online group intervention aiming to improve interoception.
  Arms: group based interoceptive intervention

SUMMARY:
Background Pulmonary hypertension is a rare and incurable condition characterised by fatigue and breathlessness. The effects of pulmonary hypertension has a significant impact on an individual's emotional wellbeing and there are currently no established psychological interventions to improve this. Interoception is defined as the ability to perceive the internal state of the body and emerging research suggests that interventions to improve interoception can improve well-being.

Aims The project aims to develop an interoceptive based intervention for those with pulmonary hypertension and examine the feasibility and acceptability of this. Additional aims are to explore the preliminary results of the intervention.

Methods A randomised control feasibility trial will be used. Thirty-two participants will be included. Participants will be patients within the Scottish Pulmonary Vascular Unit diagnosed with pulmonary hypertension and randomly assigned to either the intervention or control (waitlist) group. The intervention will be an eight-session online group and participants will complete measures for interoception, anxiety, depression, health related quality of life, as well as a feasibility and acceptability questionnaire. Quantitative analysis will include descriptive statistics and T-tests (including non-parametric versions) to analyse the feasibility and gain a preliminary understanding of the intervention.

Practical Applications It is hoped that the findings will identify a sample size for a larger trial whilst also informing future clinical practice. This project will be written up for a suitable journal and will be presented at an appropriate conference.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients under the care of the Scottish Pulmonary Vascular Unit (SPVU) at the Golden Jubilee University National Hospital (GJUNH).
* Diagnosed with any type of PH.
* Adults over 18 years.
* Fluent in English.
* Able to commit to the duration of the research (expected to be three months from initial recruitment to the end of treatment).

Exclusion Criteria:

* Individuals with current thoughts of self-harm or suicide.
* Presenting with comorbid alcohol or substance misuse.
* Currently engaging in any additional psychological interventions at the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | baseline (up to 4 weeks prior to intervention starting) and 8 weeks (during last intervention session)
  This self-report measure includes 32-items split into eight subscales of interoception. Participants rate each item on a six-point Likert scale, with higher scores indicating higher interoception. This measure has been shown to be reliable, including for those with a long-term health condition

SECONDARY OUTCOMES:
Feasibility and Acceptability Questionnaire | at 8 weeks (during last intervention session)
  A questionnaire will be developed by the lead researcher to collect information regarding feasibility and acceptability. This will be completed at the end of the intervention. Participants will be asked about different aspects of the intervention, their engagement in the study and their perceptions of change regarding managing their PH. Questionnaires will be structured statements and participants will be asked to rate their response on a five-point Likert scale. There will also be a comment section at the end of the questionnaire for participants to discuss any additional thoughts they may have.
The Generalised Anxiety Disorders Scale (GAD-7) | baseline (up to 4 weeks prior to intervention starting) and 8 weeks (during last intervention session)
  is a self-report measure that has been widely used to assess generalised anxiety within primary care settings and has shown good reliability and construct validity (Johnson et al., 2019). It consists of seven items measuring generalised anxiety and is scored on a four-point Likert scale. Scores range from 0-21 with higher scores indicating greater anxiety severity.
Patient Health Questionnaire 9 (PHQ-9) | baseline (up to 4 weeks prior to intervention starting) and 8 weeks (during last intervention session)
  a self-report measure consisting of nine items measuring depressive symptoms within primary care settings and has shown to have good psychometric properties (Johnson et al., 2019). Items are scored on a four-point Likert scale with scores ranging from 0-27, with higher scores indicating greater depression severity.
emPHasis-10 | baseline (up to 4 weeks prior to intervention starting) and 8 weeks (during last intervention session)
  a 10 item self-report questionnaire measuring HRQoL that has been specifically designed for those with PH and has been used in previous PH research (Rawling et al., 2022; Odevoglu et al., 2018). Items are scored on a six-point Likert scale with scores ranging from 0-50 with higher scores indicating lower levels of HRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Glasgow, Clydebank, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT06443580/Prot_000.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT06443580/ICF_001.pdf